CLINICAL TRIAL: NCT06583759
Title: Evaluation of Prefabricated CAD/CAM PEEK Crowns Used in Primary Molars: A Randomised Controlled Clinical Trial
Brief Title: Evaluation of Prefabricated CAD/CAM PEEK Crowns Used in Primary Molars
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Rodaina Helmy, Assistant Lecturer, Pediatric dentistry department, Faculty of dentistry, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AlexU
Record Dates: First submitted 2024-09-02; First posted 2024-09-04 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stainless Steel Crowns (Active Comparator)
  Interventions: Procedure: Full coverage Crowns
- PEEK Crowns (Experimental)
  Interventions: Procedure: Full coverage Crowns

INTERVENTIONS:
Procedure: Full coverage Crowns — The crown will be prepared accordingly. Try in of the best fitted crown will be done and cementation.

SUMMARY:
Fifty healthy cooperative children will be randomly allocated to two groups. Group I (test group) will receive CAD/CAM PEEK crowns, while group II (control group) will receive SSC. The crowns will be evaluated clinically and radiographically.

DETAILED DESCRIPTION:
A two-arm randomized controlled clinical trial. A total of 50 healthy children aged 5-7 years, will be selected from Pediatric Dentistry and Dental Public Health Department, Faculty of Dentistry, Alexandria University, Egypt. Children will be selected with scores 3 or 4 Frankl behavioral rating scale. Each child selected will have at least one mandibular second primary molar indicated for full coverage. Written informed consent will be obtained from their guardians. Participants will be randomly allocated into two groups according to the crown that will be used. Group I (test group) will receive CAD/CAM PEEK crowns, while group II (control group) will receive SSC. Using Modified Ryge's Criteria, the crowns will be examined clinically for anatomic form, restoration staining, marginal discoloration, colour match, surface roughness, marginal adaptation, proximal contact, occlusal wear of crown, wear of opposing tooth, and presence of cracks. Gingival and Plaques index scores will be recorded, as well as chairside time, patient and parental satisfaction. The patients will be recalled at 1 week then 3, 6 and 12 months for clinical follow-up. Radiographs will be taken at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Participant Inclusion Criteria

   * Age ranges from 5 - 7 years.
   * Children free of any systemic disease or special health care need (ASA I).(30)
   * Positive or definitely positive behaviour during preoperative assessments according to the Frankl Rating Scale (score 3 or 4) (Appendix I).(31)
   * Patients whose parents will give their consent to participate.
2. Tooth Inclusion Criteria

   * Mandibular second primary molars that are indicated for full coverage:(7)
   * Present opposing tooth.

Tooth Exclusion Criteria:

* Root resorption affecting more than one third of the root length.
* Clinical signs and symptoms of irreversible pulpitis or non-vitality. (Appendix II) (32)
* Fistula or abscess related to the selected tooth clinically and radiographically.
* Non restorable crowns.
* Signs of mobility or bone resorption.

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Clinical Evaluation of the crown using Modified Ryge Criteria | Day 0, 1 week , 3 months, 6 months , 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Aly Sharaf, Professor, Pediatric Dentistry, Study Director — Alexandria University
Locations (2):
- Egypt (2):
  - Faculty of Dentistry, Alexandria University, Alexandria
  - Faculty of Dentistry, Alexandria